CLINICAL TRIAL: NCT01355588
Title: A Phase 1, Double-blind, 4-way Crossover Study of the Tolerability, Safety and Pharmacokinetics of 4 Formulations of Ketorolac Tromethamine by Intranasal Administration in Healthy Volunteers
Brief Title: Tolerability, Safety and Pharmacokinetics of Four Formulations of Ketorolac Tromethamine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ROX 2005-02
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ketorolac Tromethamine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ketorolac Tromethamine (Experimental)
  Interventions: Drug: Ketorolac Tromethamine
- Ketorolac Tromethamine with 4% Lidocaine hydrochloride (HCl) (Experimental)
  Interventions: Drug: Ketorolac Tromethamine with 4% Lidocaine hydrochloride (HCl)
- Ketorolac Tromethamine with 5% Lidocaine HCl (Experimental)
  Interventions: Drug: Ketorolac Tromethamine with 5% Lidocaine HCl
- Ketorolac Tromethamine with 6% Lidocaine HCl (Experimental)
  Interventions: Drug: 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl

INTERVENTIONS:
Drug: Ketorolac Tromethamine — 30 mg Ketorolac Tromethamine intranasal (IN)
  Arms: Ketorolac Tromethamine
Drug: Ketorolac Tromethamine with 4% Lidocaine hydrochloride (HCl) — 30 mg Ketorolac Tromethamine with 4% Lidocaine HCl IN
  Arms: Ketorolac Tromethamine with 4% Lidocaine hydrochloride (HCl)
Drug: Ketorolac Tromethamine with 5% Lidocaine HCl — 30 mg Ketorolac Tromethamine with 5% Lidocaine HCl IN
  Arms: Ketorolac Tromethamine with 5% Lidocaine HCl
Drug: 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl — 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl IN
  Arms: Ketorolac Tromethamine with 6% Lidocaine HCl

SUMMARY:
This was a phase 1, double-blind, 4-way crossover study in healthy male and female volunteers. Subjects received 4 formulations of intranasal ketorolac tromethamine 30 mg. There was a wash-out period of 3-7 days between each dose. On Day 1 of each period subjects were randomised to receive either a single intranasal dose of 30 mg ketorolac tromethamine alone or single intranasal dose of 30 mg ketorolac tromethamine with 4%, 5% or 6% lidocaine hydrochloride. At the end of the study each subject had received all 4 treatments.

The primary objective of this study in healthy volunteers was to compare the safety, tolerability, and pharmacokinetics of 4 formulations of ketorolac tromethamine. A secondary objective was to monitor lidocaine hydrochloride plasma levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, aged 18 to 60 years inclusive
* Female subjects of child bearing potential must have had a negative urine pregnancy test prior to entry into the study and must not have been breast feeding
* All female subjects of child bearing potential and all male subjects with female partners of child bearing potential must have consented to use a medically acceptable method of contraception (oral or implanted contraceptive hormones, condom or diaphragm with spermicidal agent, intrauterine device or surgical sterilisation) throughout the study period
* Subject had given signed informed consent
* Subject was within 20% of normal weight for his/her height and body build according to the table of "Desirable Weights for Men and Women" (Metropolitan Life Insurance Co. 1999)
* Subject's medical history was considered normal, with no clinically significant abnormalities
* Subject was considered to be in good health in the opinion of the Investigator as determined by a pre-study physical examination with no clinically significant abnormalities, vital signs within normal range and an ECG with no clinically significant abnormalities
* Subject's pre-study clinical laboratory findings were within normal range or, if outside of the normal range, not deemed clinically significant in the opinion of the Investigator
* Subject had bilateral patent nasal airways at screening as assessed by the Investigator
* Body weight was at least 70 kg

Exclusion Criteria:

* Subject had a clinically significant illness in the 4 weeks before screening
* Use of prescribed medications in the 3 weeks prior to dosing or over-the-counter preparations for 7 days prior to dosing, except paracetamol which was allowed up to 48 hours prior to dosing. However, use of multivitamins and oral contraceptives were permitted
* Subject had a significant history of drug/solvent abuse, or a positive drugs of abuse test at screening
* Subject had history of alcohol abuse or drank in excess of 28 units per week (males) or 21 units per week (females)
* Current tobacco use or a history of smoking within the past 5 years
* Subject was, in the opinion of the Investigator, not suitable to participate in the study
* Subjects who had participated in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing
* Subjects who had a positive result of HIV screen, Hepatitis B screen or Hepatitis C screen
* Subjects with a serious adverse reaction or significant hypersensitivity to any drug
* Subjects who has donated 500 mL or more of blood within the 3 months prior to screening
* Any history of co-existing nasal polyps, NSAID sensitivity and asthma
* Allergic reaction to aspirin or other NSAIDs
* Current upper respiratory tract infection or other respiratory tract condition that could have interfered with the absorption of the nasal spray or with the assessment of AEs
* Any suspicion of rhinitis medicamentosa (chronic daily use of topical decongestants)
* Use of a monoamine oxidase inhibitor in the 14 days prior to study entry
* Active peptic ulcer disease, gastrointestinal bleeding or perforation, or a history of peptic ulcer disease or gastrointestinal bleeding
* Anemia due to unexplained or known gastrointestinal bleeding
* History of asthma or any other chronic pulmonary disorder
* Renal impairment or a risk of renal failure due to volume depletion
* Known sensitivity to lidocaine hydrochloride

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-08; Primary Completion 2005-09 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Clarke, BSc MB BS MFPM, Principal Investigator — Medeval Limited
Locations (1):
- Medeval Ltd, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 month and 2 weeks; Medeval Limited Skelton House, Manchester Science Park, Lloyd Street North, Manchester M15 6SH, U.K.
Groups:
- Treatment A, Treatment C, Treatment D, Treatment B: Treatment A: Ketorolac Tromethamine : 30 mg Ketorolac Tromethamine intranasal (IN), then; Treatment C: Ketorolac Tromethamine with 5% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 5% Lidocaine HCl IN, then; Treatment D: 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl IN, then; Treatment B: Ketorolac Tromethamine with 4% Lidocaine hydrochloride (HCl) : 30 mg Ketorolac Tromethamine with 4% Lidocaine HCl IN
- Treatment B, Treatment D, Treatment C, Treatment A: Treatment B: Ketorolac Tromethamine with 4% Lidocaine hydrochloride (HCl) : 30 mg Ketorolac Tromethamine with 4% Lidocaine HCl IN, then; Treatment D: 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl IN, then; Treatment C: Ketorolac Tromethamine with 5% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 5% Lidocaine HCl IN, then; Treatment A: Ketorolac Tromethamine : 30 mg Ketorolac Tromethamine intranasal (IN)
- Treatment C, Treatment B, Treatment A, Treatment D: Treatment C: Ketorolac Tromethamine with 5% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 5% Lidocaine HCl IN, then; Treatment B: Ketorolac Tromethamine with 4% Lidocaine hydrochloride (HCl) : 30 mg Ketorolac Tromethamine with 4% Lidocaine HCl IN, then; Treatment A: Ketorolac Tromethamine : 30 mg Ketorolac Tromethamine intranasal (IN), then; Treatment D: 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl IN
- Treatment D, Treatment A, Treatment B, Treatment C: Treatment D: 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl IN, then; Treatment A: Ketorolac Tromethamine : 30 mg Ketorolac Tromethamine intranasal (IN), then; Treatment B: Ketorolac Tromethamine with 4% Lidocaine hydrochloride (HCl) : 30 mg Ketorolac Tromethamine with 4% Lidocaine HCl IN, then; Treatment C: Ketorolac Tromethamine with 5% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 5% Lidocaine HCl IN
Period: First Intervention (Day 1)
Arm/Group | Treatment A, Treatment C, Treatment D, Treatment B | Treatment B, Treatment D, Treatment C, Treatment A | Treatment C, Treatment B, Treatment A, Treatment D | Treatment D, Treatment A, Treatment B, Treatment C
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout (3-7 Days)
Arm/Group | Treatment A, Treatment C, Treatment D, Treatment B | Treatment B, Treatment D, Treatment C, Treatment A | Treatment C, Treatment B, Treatment A, Treatment D | Treatment D, Treatment A, Treatment B, Treatment C
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (After Washout)
Arm/Group | Treatment A, Treatment C, Treatment D, Treatment B | Treatment B, Treatment D, Treatment C, Treatment A | Treatment C, Treatment B, Treatment A, Treatment D | Treatment D, Treatment A, Treatment B, Treatment C
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout (3-7 Days)
Arm/Group | Treatment A, Treatment C, Treatment D, Treatment B | Treatment B, Treatment D, Treatment C, Treatment A | Treatment C, Treatment B, Treatment A, Treatment D | Treatment D, Treatment A, Treatment B, Treatment C
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention (After Washout)
Arm/Group | Treatment A, Treatment C, Treatment D, Treatment B | Treatment B, Treatment D, Treatment C, Treatment A | Treatment C, Treatment B, Treatment A, Treatment D | Treatment D, Treatment A, Treatment B, Treatment C
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout (3-7 Days)
Arm/Group | Treatment A, Treatment C, Treatment D, Treatment B | Treatment B, Treatment D, Treatment C, Treatment A | Treatment C, Treatment B, Treatment A, Treatment D | Treatment D, Treatment A, Treatment B, Treatment C
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention (After Washout)
Arm/Group | Treatment A, Treatment C, Treatment D, Treatment B | Treatment B, Treatment D, Treatment C, Treatment A | Treatment C, Treatment B, Treatment A, Treatment D | Treatment D, Treatment A, Treatment B, Treatment C
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A, Treatment C, Treatment D, Treatment B | Treatment B, Treatment D, Treatment C, Treatment A | Treatment C, Treatment B, Treatment A, Treatment D | Treatment D, Treatment A, Treatment B, Treatment C | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 16
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.25 (17.21) | 40.75 (19.97) | 34.0 (15.90) | 50.25 (10.31) | 39.8 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 2 | 5
  Male | 2 | 4 | 3 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 4 | 4 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Anytime at pre-dose, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 15 hours (ketorolac tromethamine only), and 24 hours (ketorolac tromethamine only) post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ketorolac Tromethamine: Ketorolac Tromethamine : 30 mg Ketorolac Tromethamine intranasal (IN)
- Ketorolac Tromethamine With 4% Lidocaine Hydrochloride (HCl): Ketorolac Tromethamine with 4% Lidocaine hydrochloride (HCl) : 30 mg Ketorolac Tromethamine with 4% Lidocaine HCl IN
- Ketorolac Tromethamine With 5% Lidocaine HCl: Ketorolac Tromethamine with 5% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 5% Lidocaine HCl IN
- Ketorolac Tromethamine With 6% Lidocaine HCl: 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl : 30 mg Ketorolac Tromethamine with 6% Lidocaine HCl IN
Arm/Group | Ketorolac Tromethamine | Ketorolac Tromethamine With 4% Lidocaine Hydrochloride (HCl) | Ketorolac Tromethamine With 5% Lidocaine HCl | Ketorolac Tromethamine With 6% Lidocaine HCl
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 2059.6 (801.7) | 1963.1 (1020.8) | 1799.9 (714.1) | 2048.5 (817.6)

2. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Last Quantifiable Post-dose (AUC 0-t)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ketorolac Tromethamine | Ketorolac Tromethamine With 4% Lidocaine Hydrochloride (HCl) | Ketorolac Tromethamine With 5% Lidocaine HCl | Ketorolac Tromethamine With 6% Lidocaine HCl
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng*h/mL | 8440.6 (4021.2) | 7856.0 (4211.8) | 7561.5 (4051.2) | 8103.8 (3786.3)

3. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Infinity (AUC 0-∞)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ketorolac Tromethamine | Ketorolac Tromethamine With 4% Lidocaine Hydrochloride (HCl) | Ketorolac Tromethamine With 5% Lidocaine HCl | Ketorolac Tromethamine With 6% Lidocaine HCl
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng*h/mL | 9061.9 (4526.8) | 8694.5 (4477.1) | 8086.8 (4608.2) | 8677.6 (4301.0)

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Ketorolac Tromethamine | Ketorolac Tromethamine With 4% Lidocaine Hydrochloride (HCl) | Ketorolac Tromethamine With 5% Lidocaine HCl | Ketorolac Tromethamine With 6% Lidocaine HCl
Number analyzed (Participants) | 16 | 16 | 16 | 16
hours | 0.510 [0.50 to 1.50] | 0.500 [0.25 to 4.00] | 0.390 [0.25 to 0.75] | 0.410 [0.25 to 0.50]

ADVERSE EVENTS:
Time Frame: 1 month and 2 weeks
Arm/Group | Ketorolac Tromethamine | Ketorolac Tromethamine With 4% Lidocaine Hydrochloride (HCl) | Ketorolac Tromethamine With 5% Lidocaine HCl | Ketorolac Tromethamine With 6% Lidocaine HCl
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 11/16 | 9/16 | 9/16 | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketorolac Tromethamine (N=16) | Ketorolac Tromethamine With 4% Lidocaine Hydrochloride (HCl) (N=16) | Ketorolac Tromethamine With 5% Lidocaine HCl (N=16) | Ketorolac Tromethamine With 6% Lidocaine HCl (N=16)
Fatigue (General disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 6 | 6
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 6 | 3
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No